CLINICAL TRIAL: NCT05898009
Title: Contribution of Oncogenetics in Breast Cancer in Reunion Epidemiology of Breast Cancer in Reunion: Study of the Reunion Mutation on BRCA2
Acronym: CanSeR-OGen
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023/CHU/04
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Genetic Disease; BRCA2 Mutation
Keywords: reunion
MeSH Terms: conditions — Breast Neoplasms; Genetic Diseases, Inborn | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BRCA2 mutation detection (Experimental)
  Interventions: Genetic: blood sample for BRCA2 mutation detection

INTERVENTIONS:
Genetic: blood sample for BRCA2 mutation detection — blood sample

SUMMARY:
In mainland France, breast cancer is the most common cancer in women, with an estimated incidence of over 58,000 new cases. Even if breast cancer is a cancer with a good prognosis, it is responsible for more than 12,000 deaths per year (first cause of death by cancer in women in France).

Breast cancer is a multifactorial disease, which results from the interaction between environmental, lifestyle, hormonal and genetic risk factors.

In Reunion, more than 400 cases of breast cancer are diagnosed annually. As in mainland France, it is by far the most common cancer in Reunionese women, and its incidence continues to increase significantly since the age-standardized incidence rate increased by 28% between 2007 and 2017 to establish at 64.2/100,000 AP.

Two studies carried out in patients carrying mutations in the breast-ovary predisposition genes in Reunion, showed that more than 50% of patients carrying BRCA mutation have a mutation specific to the Reunion population on the BRCA2 gene.

These two studies, which confirm the genetic specificities of Reunion already described in other pathologies (Mucoviscidosis or Friedreich's Ataxia), suggest that this mutation could have a significant frequency in patients with breast cancer. Thus, evaluating the prevalence of this mutation in patients with breast cancer in Réunion would make it possible to adapt the indications for access to the oncogenetics consultation and the associated preventive measures

ELIGIBILITY:
Inclusion Criteria:

* Domiciled in Reunion at the time of the diagnosis
* Who is diagnosed with a first breast cancer (in situ or invasive) confirmed by anatomopathological examination during the inclusion period Or Who is diagnosed with a second breast cancer (in situ or invasive) confirmed by pathological examination during the inclusion period, contralateral to the first or at least 5 years after remission of the first
* Having agreed to participate in the study;
* Affiliates or beneficiaries of a social security scheme

Exclusion Criteria:

* Carriers of breast lymphoma,
* Minor patients or patients under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2025-03-22 (Estimated); Study Completion 2026-03-22 (Estimated)

PRIMARY OUTCOMES:
determine the prevalence of the Réunion mutation in the BRCA2 gene (c.2612C>A mutation of exon 11) in the population of individuals residing in Réunion who are diagnosed with breast cancer. | inclusion day

CONTACTS AND LOCATIONS:
Locations (1):
- Mireille IRABE, Saint-Pierre, France

IPD SHARING:
Plan to Share IPD: No